CLINICAL TRIAL: NCT04824950
Title: Circulating Tumor DNA in Primary Mediastinal Large B-cell Lymphoma (PMBL)
Acronym: CAMIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB20.03
Record Dates: First submitted 2021-03-23; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Primary Mediastinal Large B-cell Lymphoma
Keywords: Primary Mediastinal Large B-cell Lymphoma; Circulating tumor DNA; Next Generation sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monitoring of Circulating Tumor DNA (Other)
  Interventions: Other: Circulating tumor DNA monitoring

INTERVENTIONS:
Other: Circulating tumor DNA monitoring — Monitoring of circulating tumor DNA after 2 and 4 cycles of chemotherapy

SUMMARY:
The purpose of this study is to compare the predictive value in terms of specificity of circulating tumor DNA (ctDNA) and positron emission computed tomography (PET-CT) after 2 cycles of chemotherapy (C2), on the probability of obtaining a metabolic complete response after 4 cycles of induction chemotherapy (C4) in patients with primary mediastinal large B cell lymphoma (PMBL) receiving standard R-CHOP14 or R-ACVBP.

DETAILED DESCRIPTION:
The majority of studies with PMBL patients pinpoint the importance of being able to identify primary chemo refractory patients at an early stage, in order to be able to improve their prognosis. Indeed, a biomarker such as circulating tumor DNA (ctDNA) monitoring would be of great help to better assess the therapeutic response and offer an individualized care given the frequent positive residual uptake of the mediastinum at end of treatment. Indeed, ctDNA can be detected with Next-Generation Sequencing (NGS).

The hypothesis of this study is that it would be helpful to prospectively compare the predictive value of ctDNA versus PET on the capacity to detect primary refractory patients after 2 or 4 cycles of first line chemotherapy.

To date, there are no prospective studies reporting the evolution of the tumor clone under treatment or after obtaining complete remission in PMBL. The establishment of this prospective, multicenter, ambitious and original pilot project will make it possible to structure the analysis of tumor DNA circulating within these centers caring for patients with lymphomas within LYSA group.

The notion of minimal residual disease (MRD) has shown its interest in follicular lymphomas and mantle cell lymphomas. The level of sensitivity of NGS-type approaches on the one hand and the informativeness of the recurrent mutations recently described on the other hand constitute two elements for reconsidering the problem of MRD in PMBLs. Molecular MRD by analysis of circulating tumor DNA could constitute a new marker for monitoring response to treatment in addition to PET-CT and be useful as a tool for non-invasive tumor sequencing at diagnosis and at relapse, in order to to determine the eligibility for possible targeted therapies (based on the inactivation of mutated genes) or immunotherapies.

This study will evaluate the prognostic value of obtaining a quantified complete molecular response (RMC) by analysis of free circulating DNA (ctDNA) after 2 and 4 cycles of first-line chemotherapy (C2 and C4) for the treatment of PMBL, and that of positron emission computed tomography (PET) performed at the same time, on overall survival and progression-free survival.

The investigators will describe 3 different populations of patients included in the study:

1. Patients with "negative" plasma DNA at diagnosis (defined by the absence of somatic mutation detectable at diagnosis by ctDNA analysis)
2. Patients with "positive" plasma DNA at diagnosis (defined by the presence of at least one somatic mutation detectable at diagnosis by ctDNA analysis) and whose plasma DNA becomes "negative" after 2 cycles of chemotherapy
3. Patients with "positive" plasma DNA and whose plasma DNA remains "positive" after 2 cycles of chemotherapy For these 3 patient profiles, we will perform comparisons, search for correlations with different variables and perform univariate and multivariate statistical analyzes.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age,
* Suffering from a diffuse primary B lymphoma of the mediastinum, newly diagnosed locally on a biopsy with anatomopathological analysis according to the recommendations of the WHO 2016 classification of hematological malignancies,
* All stages (I-IV)
* All IPI scores (0-5)
* With mediastinal involvement,
* Untreated (apart from emergency corticosteroid therapy less than 2mg/kg/day for 7 days),
* Treatment with R-CHOP-14 or R-ACVBP with PET-CT guided strategy (delta SUVmax) to be initiated,
* Tumor fixation above liver background on pre-treatment FDG PET/CT/CT (Deauville score ≥4),
* Having signed the informed consent prior to any study procedure
* Affiliated or beneficiary of a social protection plan.

Exclusion Criteria:

* Patient who has already started chemotherapy treatment,
* Contraindication to FDG PET-CT,
* No mediastinal involvement,
* Positive HIV serology,
* Positive hepatitis B or C serology with positive viral load,
* Protected adult (under guardianship or curatorship),
* Pregnant or breastfeeding women,
* Patient unable to understand the study for any reason or to comply with the constraints of the trial (language, psychological, geographical problems, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2021-03-22 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between circulating tumoral DNA detection and complete molecular response | 4 months
  specificity of ctDNA at Cycle 2 of chemotherapy on the prediction of achieving a complete metabolic response (determined by PET-CT scan) at cycle 4 of chemotherapy

SECONDARY OUTCOMES:
Evaluation of complete metabolic response | at the end of first line treatment
  Proportion of patient in complete metabolic response at the end of first line treatment
Evaluation of response | At the end of 4 cycles of chemotherapy
  Percentage of patients in complete metabolic response, partial metabolic response, stable disease or pregression after 4 cycles of chemotherapy
Evaluation of response | At the end of treatment
  Percentage of patients in complete metabolic response, partial metabolic response, stable disease or pregression at the end of treatment
overall survival | 3 years
  Time between death and inclusion
Event free survival | 3 years
  Lenght of time after the end of tratment and events like progression, lake of response, relapse of death whatever the cause
genic expression profile | 3 years
  Next-Generation-sequencing on diagnostic biopsy
Genomic sequencing of circulating tumor DNA | 3 years
  Determination of molecular profile and evaluation of pronostic impact
Correlation between Next-Generation-Sequencing on tumor and molecular profile obtained on circulating tumor DNA | 3 years
  Comparison between the result of Next generation Sequencing and the molocular profile obtained on circulation tumor DNA of each patient

CONTACTS AND LOCATIONS:
Overall Officials: VINCENT CAMUS, MD, Principal Investigator — Centre Henri Becquerel; PIERRE SESQUES, MD, Principal Investigator — Centre Hospitalier Lyon Sud
Locations (2):
- France (2):
  - Centre Hospitalier Lyon Sud, Lyon
  - Centre Henri Becquerel, Rouen